CLINICAL TRIAL: NCT00004935
Title: Randomized Phase III Trial of Herceptin® Followed by Chemotherapy Plus Herceptin® Versus the Combination of Herceptin® and Chemotherapy as Palliative Treatment in Patients With HER2- Overexpressing Advanced/Metastatic Breast Cancer.
Brief Title: Herceptin Followed by Chemotherapy in Treating Women With Metastatic Breast Cancer That Overexpresses HER2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Trial is Life long follow-up: to reduce ressources and costs - trial terminated prematurely.
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 22/99; SWS-SAKK-22/99 (Other: SAKK); EU-99028 (Other: SAKK)
Record Dates: First submitted 2000-03-07; First posted 2003-01-27 (Estimated); Last update posted 2023-04-18 (Actual); Status verified 2022-03

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Herceptin™ (Her) (Active Comparator): Herceptin™ (Her) loading dose 4 mg/kg iv, followed by 2 mg/kg iv weekly or loading dose 8 mg/kg iv, followed by 6 mg/kg iv every 3 weeks; at time of progression add chemotherapy
  Interventions: Drug: Herceptin™ (Her)
- Herceptin™+Chemo (Active Comparator): Herceptin™ (Her) loading dose 4 mg/kg iv, followed by 2 mg/kg iv weekly or loading dose 8 mg/kg iv, followed by 6 mg/kg iv every 3 weeks, and chemotherapy
  Interventions: Drug: Herceptin™ (Her) + chemo

INTERVENTIONS:
Drug: Herceptin™ (Her) — Herceptin™ (Her) loading dose 4 mg/kg iv, followed by 2 mg/kg iv weekly or loading dose 8 mg/kg iv, followed by 6 mg/kg iv every 3 weeks; at time of progression add chemotherapy
  Arms: Herceptin™ (Her)
Drug: Herceptin™ (Her) + chemo — Herceptin™ (Her) loading dose 4 mg/kg iv, followed by 2 mg/kg iv weekly or loading dose 8 mg/kg iv, followed by 6 mg/kg iv every 3 weeks, and chemotherapy
  Arms: Herceptin™+Chemo

SUMMARY:
RATIONALE: To compare efficacy, toxicity and quality of life of the sequential administration of Her alone followed, at PD, by the combination with Chemotherapy (Arm A) vs. the upfront combination of Her and Chemotherapy (Arm B) in patients with advanced/metastatic breast cancer.

PURPOSE: Trial SAKK 22/99 addresses clinically relevant and currently unresolved questions regarding the optimal use of Herceptin in the treatment of patients with advanced/metastatic breast cancer.

DETAILED DESCRIPTION:
In advanced HER2+ breast cancer the impact of combining Trastuzumab (T) and chemotherapy (chemo) versus T alone followed by the addition of chemo at disease progression has not been properly studied.

The trial compared efficacy, toxicity and quality of life of sequential administration of T followed, at progression, by combination with chemo (T>TChemo) versus the upfront combination of T and chemo (TChemo) in patients with HER2+ advanced breast cancer.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed HER2-overexpressing metastatic breast carcinoma
* Clinically or radiologically measurable or evaluable disease

  * Bidimensionally or unidimensionally measurable lesions
* No ascitic, pleural, or pericardial effusions, osteoblastic bone metastases, or carcinomatous lymphangitis of the lung as only indicator lesion
* No known clinical brain or meningeal involvement
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 to 70

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* ECOG 0-1 OR
* SAKK 0-1

Life expectancy:

* At least 12 weeks

Hematopoietic:

* Hemoglobin at least 10 g/dL
* Platelet count at least 100,000/mm^3
* Absolute neutrophil count at least 2,000/mm^3

Hepatic:

* Bilirubin normal
* SGOT and/or SGPT no greater than 2 times upper limit of normal (ULN) (3 times ULN if proven liver metastases) OR
* No SGOT and/or SGPT greater than 1.5 times ULN if alkaline phosphatase greater than 2.5 times ULN

Renal:

* Creatinine no greater than 1.25 times ULN

Cardiovascular:

* LVEF normal
* No history of atrial ventricular arrhythmia, congestive heart failure, or angina pectoris, even if medically controlled
* No history of second or third-degree heart blocks
* No uncontrolled hypertension

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No pre-existing motor or sensory neuropathy grade 2 or greater
* No psychiatric disorder that would preclude informed consent
* No other prior malignancy except curatively treated nonmelanoma skin cancer or carcinoma in situ of the cervix
* No definite contraindications for use of corticosteroids
* No other concurrent serious illness or medical condition

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Prior adjuvant or neoadjuvant chemotherapy allowed
* No more than 2 prior chemotherapy regimens for metastatic disease
* No prior cumulative dose of doxorubicin greater than 240 mg/m^2
* No prior cumulative dose of epirubicin greater than 360 mg/m^2
* No prior taxanes

Endocrine therapy:

* Prior hormonal therapy as adjuvant treatment or for metastatic disease allowed
* No concurrent corticosteroids unless started more than 6 months prior to study and at low doses (i.e., no greater than 20 mg methylprednisolone or equivalent)

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* No other concurrent anticancer drugs
* No other concurrent experimental drugs
* No concurrent bisphosphonates unless initiated more than 3 months prior to study

  * Chronic use allowed provided bone metastases are not sole indicator lesions

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 1999-08-30 (Actual); Primary Completion 2014-11-06 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Time to progression on combined HerChemo (TTPHerChemo) | 8 weeks

SECONDARY OUTCOMES:
Response rate | 8 weeks
Time to first progression | 8 weeks
Time to treatment failure | 8 weeks
Overall survival | 8 weeks
Adverse events | 8 weeks
Predictive value of serum HER2/neu ECD levels on clinical outcome | 8 weeks
Conversion rate of estrogen receptor status | 8 weeks
Association of immunoprofiles of erbB-1, erbB-2, erbB-3 and erbB-4 with clinical outcome | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pagani Olivia, MD, Study Chair — Istituto Oncologico della Svizzera Italiana IOSI
Locations (17):
- Italy (2):
  - European Institute of Oncology, Milan
  - Ospedale di Circolo e Fondazione Macchi, Varese
- Switzerland (15):
  - Kantonsspital Aarau, Aarau
  - Kantonsspital Baden, Baden
  - Universitaetsspital-Basel, Basel
  - Istituto Oncologico della Svizzera Italiana - Ospedale Regionale Bellinzona e Valli, Bellinzona
  - Inselspital Bern, Bern
  - Kantonsspital Graubuenden, Chur
  - Hopital Cantonal Universitaire de Geneve, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Ospedale Regionale di Lugano, Lugano
  - Praxis Dr. Beretta, Rheinfelden
  - Kantonsspital - St. Gallen, Sankt Gallen
  - Regionalspital, Thun
  - Onkozentrum, Zurich
  - City Hospital Triemli, Zurich
  - UniversitaetsSpital Zuerich, Zurich

REFERENCES:
- [Derived] Eppenberger-Castori S, Klingbiel D, Ruhstaller T, Dietrich D, Rufle DA, Rothgiesser K, Pagani O, Thurlimann B. Plasma HER2ECD a promising test for patient prognosis and prediction of response in HER2 positive breast cancer: results of a randomized study - SAKK 22/99. BMC Cancer. 2020 Feb 11;20(1):114. doi: 10.1186/s12885-020-6594-0. PMID 32046665
- [Derived] Schmid S, Klingbiel D, Aebi S, Goldhirsch A, Mamot C, Munzone E, Nole F, Oehlschlegel C, Pagani O, Pestalozzi B, Rochlitz C, Thurlimann B, von Moos R, Weder P, Zaman K, Ruhstaller T. Long-term responders to trastuzumab monotherapy in first-line HER-2+ advanced breast cancer: characteristics and survival data. BMC Cancer. 2019 Sep 10;19(1):902. doi: 10.1186/s12885-019-6105-3. PMID 31500588